CLINICAL TRIAL: NCT04046731
Title: The Negative Predictive Value and Non-irritant Skin Testing Concentrations of Neuromuscular Blocking Agents Utilized During Perioperative Hypersensitivity Evaluation
Brief Title: Neuromuscular Blocking Agents Utilized During Perioperative Hypersensitivity Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexei Gonzalez-Estrada, MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-007462
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): Study team is developing a new diagnostic skin testing procedure for patients who receive NMBAs during surgery in order to determine Negative Predictive Values and Non-Irritant Concentrations.
  Interventions: Diagnostic Test: Skin Testing

INTERVENTIONS:
Diagnostic Test: Skin Testing — Percutaneous skin prick followed by Intradermal Injections of NMBAs at increasing concentrations compared with an established positive and negative control.

SUMMARY:
The researchers are trying to develop an allergy skin test to help predict allergic responses to medications commonly given to patients during surgery.

DETAILED DESCRIPTION:
This study will be a prospective study to accurately determine the negative predictive value of skin testing with NMBAs.

It is hypothesized that the concentrations that should be used for NMBAs are actually much lower than previously recommended and that the higher incidence of identifiable NMBA induced allergic reactions during anesthesia in the past may be due to irritation of the skin rather than a true allergic reaction (false positives).

ELIGIBILITY:
Inclusion Criteria:

* All adults > or = to 18 y/o undergoing surgery

Exclusion Criteria:

* Minors under the age of 18 y/o, Adults unable to consent, or those Adults with previous allergic reaction history during previous surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Non-Irritant Concentrations to common NMBAs | 1 Year
  Determine the NIC to common NMBAs

SECONDARY OUTCOMES:
Negative Predictive Value of Intradermal Skin Testing to commonly used NMBAs | 1 Year
  Determine Negative Predictive Value of Intradermal Skin Testing to commonly used NMBAs
Max Concentration used when skin testing to NMBAs | 1 Year
  Close gap on the variability of the maximal concentration used when skin testing NMBAs.

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Gonzalez Estrada, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials